CLINICAL TRIAL: NCT04304976
Title: Clinical Trial ROBERT® - Project Active Training
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Lifescience-Robotics (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: N-20190038
Record Dates: First submitted 2020-02-26; First posted 2020-03-12 (Actual); Last update posted 2021-02-21 (Actual); Status verified 2020-03

CONDITIONS: Apoplexy; Stroke; Spinal Cord Injuries; Safety; Usability
MeSH Terms: conditions — Stroke; Spinal Cord Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Training with ROBERT® Passive (Experimental): Training performed with ROBERT® in passive mode, resulting in active assistive training.
  Interventions: Device: ROBERT®
- Training with ROBERT® Active (Experimental): Traning performed with ROBERT® in Active mode, resulting in active resistive training.
  Interventions: Device: ROBERT®

INTERVENTIONS:
Device: ROBERT® — Robotic Rehabilitation intervention ROBERT®, designed for early, and supplementary therapy of patients.

SUMMARY:
The overall purpose with this clinical trial is to, monitor and secure ROBERT®'s clinical performance and safety in a clinical environment in the regional hospital North Denmark, Neuro Unit North. The purpose of the study is to investigate if ROBERT® has the ability to 1. Perform guided active training. 2. Perform resistance based active training. And validate the safety of ROBERT® in a clinical environment.

ELIGIBILITY:
Inclusion Criteria:

* Hospitalised patients at Neuro Unit North, during the trial period.
* 18 years or older.
* Can read, understand and speak Danish
* Reduced motor function in lower extremities.

Exclusion Criteria:

* No able to sign informed consent.
* Cannot read, understand or speak Danish
* Patients with unstable fractures in columna, pelvis or lower extremities.
* Patients with the risk of ulcers, or with exceedingly sensitive skin.
* The patient is refusing to train with ROBERT®

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2019-11-27 (Actual); Primary Completion 2020-01-16 (Actual); Study Completion 2020-04-21 (Actual)

PRIMARY OUTCOMES:
Active training and assistive training capabilities (3 active and 3 passive motions): evaluated as passed/not passed | Up to 19 weeks
  1. Active training capabilities will be assessed, 3 active motions are planned (the therapist has to be active) by the therapist, and manually performed by hand. The resistance perceived by the therapist is then compared to the expert opinion of the therapist to evaluate if this correlates with, small, medium, and large resistance. This is evaluated as passed/not passed for all 3 motions
  2. Active assistive training capabilities will be assessed: 3 passive motions are planned (the robot moves, the therapist follows movement), by the therapist and the robot starts performing the motions, the therapist performs a small, moderate and large assistive movement in conjunction with the robot. The results in % of activity in the path of motion are displayed, and the therapist evaluates if this is in agreement with what they would categorise as a small, moderate and large assistive movement respectively. This is evaluated as passed/not passed for all 3 motions.
Safety, Capture adverse events. | Up to 19 weeks
  Safety is evaluated during patient use, nr of treatment-related adverse events is recorded during training sessions.

CONTACTS AND LOCATIONS:
Overall Officials: Helle Rovsing Jørgensen, Therapist, Principal Investigator — Neuro Unit Nord, Denmark
Locations (1):
- Region Hospital, Neuro Unit Nord., Frederikshavn, North Denmark, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Wunsch H, Guerra C, Barnato AE, Angus DC, Li G, Linde-Zwirble WT. Three-year outcomes for Medicare beneficiaries who survive intensive care. JAMA. 2010 Mar 3;303(9):849-56. doi: 10.1001/jama.2010.216. PMID 20197531
- [Background] Needham DM, Davidson J, Cohen H, Hopkins RO, Weinert C, Wunsch H, Zawistowski C, Bemis-Dougherty A, Berney SC, Bienvenu OJ, Brady SL, Brodsky MB, Denehy L, Elliott D, Flatley C, Harabin AL, Jones C, Louis D, Meltzer W, Muldoon SR, Palmer JB, Perme C, Robinson M, Schmidt DM, Scruth E, Spill GR, Storey CP, Render M, Votto J, Harvey MA. Improving long-term outcomes after discharge from intensive care unit: report from a stakeholders' conference. Crit Care Med. 2012 Feb;40(2):502-9. doi: 10.1097/CCM.0b013e318232da75. PMID 21946660
- [Background] I. Com, Global strategy and action plan on ageing and health. 2017.
- [Background] "NEUROLOGICAL DISORDERS public health challenges WHO Library Cataloguing-in-Publication Data," 2006.
- [Background] Wist S, Clivaz J, Sattelmayer M. Muscle strengthening for hemiparesis after stroke: A meta-analysis. Ann Phys Rehabil Med. 2016 Apr;59(2):114-24. doi: 10.1016/j.rehab.2016.02.001. Epub 2016 Mar 8. PMID 26969343
- [Background] English C, Bernhardt J, Crotty M, Esterman A, Segal L, Hillier S. Circuit class therapy or seven-day week therapy for increasing rehabilitation intensity of therapy after stroke (CIRCIT): a randomized controlled trial. Int J Stroke. 2015 Jun;10(4):594-602. doi: 10.1111/ijs.12470. Epub 2015 Mar 19. PMID 25790018
- [Background] Sarkies MN, White J, Henderson K, Haas R, Bowles J; Evidence Translation in Allied Health (EviTAH) Group. Additional weekend allied health services reduce length of stay in subacute rehabilitation wards but their effectiveness and cost-effectiveness are unclear in acute general medical and surgical hospital wards: a systematic review. J Physiother. 2018 Jul;64(3):142-158. doi: 10.1016/j.jphys.2018.05.004. Epub 2018 Jun 19. PMID 29929739
- [Background] Peiris CL, Taylor NF, Shields N. Extra physical therapy reduces patient length of stay and improves functional outcomes and quality of life in people with acute or subacute conditions: a systematic review. Arch Phys Med Rehabil. 2011 Sep;92(9):1490-500. doi: 10.1016/j.apmr.2011.04.005. PMID 21878220
- [Background] Peiris CL, Shields N, Brusco NK, Watts JJ, Taylor NF. Additional Physical Therapy Services Reduce Length of Stay and Improve Health Outcomes in People With Acute and Subacute Conditions: An Updated Systematic Review and Meta-Analysis. Arch Phys Med Rehabil. 2018 Nov;99(11):2299-2312. doi: 10.1016/j.apmr.2018.03.005. Epub 2018 Apr 7. PMID 29634915
- [Background] Lohse KR, Lang CE, Boyd LA. Is more better? Using metadata to explore dose-response relationships in stroke rehabilitation. Stroke. 2014 Jul;45(7):2053-8. doi: 10.1161/STROKEAHA.114.004695. Epub 2014 May 27. PMID 24867924
- [Background] Lang CE, Lohse KR, Birkenmeier RL. Dose and timing in neurorehabilitation: prescribing motor therapy after stroke. Curr Opin Neurol. 2015 Dec;28(6):549-55. doi: 10.1097/WCO.0000000000000256. PMID 26402404
- [Background] "Ét sikkert og sammenhaengende sundhedsnetvaerk for alle."
- [Background] Masiero S, Poli P, Rosati G, Zanotto D, Iosa M, Paolucci S, Morone G. The value of robotic systems in stroke rehabilitation. Expert Rev Med Devices. 2014 Mar;11(2):187-98. doi: 10.1586/17434440.2014.882766. Epub 2014 Jan 30. PMID 24479445
- [Background] Semprini M, Laffranchi M, Sanguineti V, Avanzino L, De Icco R, De Michieli L, Chiappalone M. Technological Approaches for Neurorehabilitation: From Robotic Devices to Brain Stimulation and Beyond. Front Neurol. 2018 Apr 9;9:212. doi: 10.3389/fneur.2018.00212. eCollection 2018. PMID 29686644
- [Background] Langhorne P, Coupar F, Pollock A. Motor recovery after stroke: a systematic review. Lancet Neurol. 2009 Aug;8(8):741-54. doi: 10.1016/S1474-4422(09)70150-4. PMID 19608100